CLINICAL TRIAL: NCT02911129
Title: Effects of Prism Adaption and rTMS on Brain Connectivity and Visual Representation
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 160170; 16-N-0170
Record Dates: First submitted 2016-09-21; First posted 2016-09-22 (Estimated); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Normal Physiology; Stroke
Keywords: Chronic Stroke; Neglect; Transcranial Magnetic Stimulation; Visual and Motor Integration; Visual Fields; Natural History
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteer: Inclusion Criteria for Healthy Volunteers/Age-matched Controls
- Patients: Patients with neglect after a right hemisphere brain lesion

SUMMARY:
Background:

After a stroke, the balance between the two halves of the brain can be lost. This may cause people to lose the ability to perceive a side of space. This is called neglect. Having people wear prism glasses (called PA) can reduce neglect symptoms. Researchers want to find out more about how PA, and whether it restores the balance in the brain.

Objective:

To learn how prism adaption temporarily changes vision and connections in the brain.

Eligibility:

People ages 18 75 with brain damage of the right side of the brain from a stroke or other cause, leading to neglect.

Healthy volunteers ages 18 75.

Design:

Participants will have 1 3 visits.

Participants will be screened with a neurological exam. They may also have:

Tests of thinking and vision

Tests to see which eye and hand they prefer

A pregnancy test

All participants will:

Answer questions about their personality, style of thinking, and beliefs.

Do simple tasks on paper or computer

Have magnetic resonance imaging. They will lie on a table that can slide in and out of a cylinder in a strong magnetic field. Participants will lie still or do computer tasks in the scanner.

Participants may also have:

Transcranial magnetic stimulation. A brief electrical current passes through a wire coil on the scalp. This creates a magnetic pulse that affects brain activity. Participants may be asked to tense certain muscles or perform simple actions or tasks.

PA. They will sit in front of a board and point to a dot on it while they wear prism glasses that shift vision to the left or right....

DETAILED DESCRIPTION:
OBJECTIVES:

The ability to efficiently select information from the environment relies on a balanced interaction between the right and left hemispheres. Hemispatial neglect, most frequently following damage to the right hemisphere, has been hypothesized to result from the breakdown of this interhemispheric balance. There is evidence from transcranial stimulation studies that the breakdown of this interhemispheric balance is reflected in fronto-parietal connectivity. The primary goal of this study is to test whether altering the balance between the left and right hemispheres, with repetitive transcranial magnetic stimulation (rTMS) or prism adaptation (PA), will affect functional connectivity measured with functional magnetic resonance imaging (fMRI). We will also explore the relationship between the changes in functional connectivity and behavioral performances.

STUDY POPULATION: Healthy adult volunteers and patients with neglect after a right hemisphere damage.

DESIGN: The study contains three experiments. Experiment 1 is designed to investigate the mechanism of the changes induced by PA in both resting state functional connectivity in neglect patients and healthy volunteers (a two-arm parallel study). Experiment 2 is designed to investigate the mechanism of the changes in resting state functional connectivity induced by lPA, rPA, nPA in healthy volunteers with right dominant eyes and lPA in healthy volunteer with left dominant eye (a four-arm parallel study). Experiment 3 is designed to see if inhibitory rTMS over the right posterior parietal cortex (PPC) can influence functional connectivity and visuospatial bias in healthy volunteers (a crossover study).

OUTCOME MEASURES: For all three experiments the primary outcome measure is the change (or difference) in fronto-parietal resting state connectivity between post and pre PA or rTMS procedure. The secondary outcome measures are the changes in visual field representation and in visuo-motor and cognitive behavior accompanying these manipulations.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion Criteria for all participants:

All participants must have had a neurological examination by a NINDS physician within the last two years, a clinical MRI within the last year, and be able to read, write and speak English.

Experiment 2 requires 63 healthy volunteers having right dominant eye and 21 volunteers having left dominant eye. Therefore, healthy volunteers with left dominant eye will be recruited until the necessary number is reached. We estimate we will have to screen 150

healthy volunteers. Participants for whom the study was not completed due to technical problems and who did not undergo prism adaptation or TMS will be retested and data from the incomplete session will not be analyzed.

A-Inclusion Criteria for Healthy volunteers/Age-matched Controls

Experiment 1

* Age 18-75 (inclusive; we will try to match this to the stroke group)
* Montreal Cognitive Assessment score greater than or equal to 26
* Absence of neglect at time of testing (Diller test score less than or equal to 2)

Experiments 2 and 3

* Right-handedness
* Age 18-35 (inclusive)
* Twelve or more years of education
* Are able to see a dot of size 0.2 inches at a distance of 22.5 inches without glasses or with contact lenses (only for Experiment 2)

B-Inclusion Criteria for Patients

Experiment 1

* Age 18-75 (inclusive)
* Montreal Cognitive Assessment score greater than or equal to 26
* A right hemisphere stroke or other focal, non-progressive, brain lesion resulting in neglect
* Minimum of 30 days from lesion onset to testing
* Evidence of neglect at time of testing (Diller test score greater than or equal to 5)

EXCLUSION CRITERIA:

A- Exclusion Criteria for Healthy volunteers

* Significant illness affecting the central nervous system
* History of seizure (for Experiment 3)
* Inability to give informed consent
* Concurrent use of sedating medications
* Trained to write in other than left to right direction
* Ferromagnetic metal in the cranial cavity or eye, e.g. aneurysm clip, implanted neural stimulator, cochlear implant, or ocular foreign body
* Implanted cardiac pacemaker or auto-defibrillator or pump
* Non-removable body piercing
* Claustrophobia
* Inability to lie supine for 1.5 hour
* Pregnancy
* Members of the NINDS Behavioral Neurology Unit (BNU)

B- Exclusion Criteria for Patients and Age-matched Controls:

* Significant illness affecting the central nervous system, other than right hemisphere lesion causing neglect in patients
* Inability to give informed consent
* Concurrent use of sedating medications
* Ferromagnetic metal in the cranial cavity or eye, e.g. aneurysm clip, implanted neural stimulator, cochlear implant, or ocular foreign body
* Implanted cardiac pacemaker or auto-defibrillator or pump
* Non-removable body piercing
* Claustrophobia
* Inability to lie supine for 1.5 hour
* Pregnancy
* Members of the NINDS Behavioral Neurology Unit (BNU)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary Clinical
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2016-11-04 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Experiment 1: The primary outcome measure will be the change in the strength of the fronto-parietal resting state network (RSN) after rPA in neglect patients. | 1 week
  Measurement of Change
Experiments 2: The primary outcome measure will be the change in the strength of the fronto-parietal resting state network (RSN) after rPA or lPA or nPA. | 1 week
  Measurement of change
Experiment 3: The primary outcome measure will be the change in the strength of the fronto-parietal resting state network (RSN) after cTBS over the PPC versus cTBS over the vertex. | 3 weeks
  Measurement of change

SECONDARY OUTCOMES:
Experiment 1: The change of preferred center and size in the different region of interest (ROI) in the parietal cortex, and the change in open loop pointing task performances after rPA. | 1 week
  Observation of changeExperiment 1: The change of preferred center (visual field location) and size (visual field extent) (i.e. population receptive field) in the different region of interest (ROI) in the parietal cortex, and the change in open loop pointing task performances after rPA.
Experiments 2: The change of preferred center and sizein the different region of interest (ROI) in the parietal cortex, and the change in open loop pointing task performances after rPA or lPA, or nPA | 1 week
  Observation of changeExperiments 2: The change of preferred center (visual field location) and size (visual field extent) (i.e. population receptive field) in the different region of interest (ROI) in the parietal cortex, and the change in open loop pointing task performances after rPA or lPA, or nPA
Experiments 3: The change in perceptual line bisection performances after r cTBS over PPC or cTBS over the vertex. | 1 week
  Oberservation of change

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Wassermann, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-N-0170.html